CLINICAL TRIAL: NCT06289062
Title: Neoadjuvant Chemotherapy Plus Camrelizumab (NACI Therapy) for Fertility Preservation in FIGO Stage IB1 Cervical Cancer
Brief Title: Neoadjuvant Chemotherapy Plus Camrelizumab for FIGO Stage IB1 Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Third Military Medical University (Other); Beijing Friendship Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Tianjin Medical University (Other); West China Second University Hospital (Other); Xiangya Hospital of Central South University (Other); Qilu Hospital of Shandong University (Other); Gansu Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Shengjing Hospital (Other); Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Kezhen Li, Prof, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NACI-CERV-005
Record Dates: First submitted 2024-02-19; First posted 2024-03-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancer; Neoadjuvant Chemoimmunotherapy; Fertility Preservation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; Cisplatin; Taxes; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NACI in FIGO ⅠB1 Cervical Cancer (Experimental): Neoadjuvant chemotherapy plus camrelizumab for ⅠB1 Cervical Cancer. Patients first received one cycle of platinum-based doublet priming chemotherapy. After 3 weeks, participants subsequently received two cycles of the PD-1 inhibitor camrelizumab combined with chemotherapy every 3 weeks. The study will be conducted in two stages: (1) Patients enrolled in the first stage with tumors ≤2 cm and no new lesions after completion of treatment will undergo cone biopsy + pelvic lymphadenectomy or SLN mapping. Those who meet ConCerv criteria will undergo a second TCT, human papillomavirus (HPV) and colposcope 3 months later, and those who do not meet ConCerV criteria will undergo radical cervical surgery. (2) Patients enrolled in the second stage with tumors ≤2 cm and no new lesions underwent cervical biopsy + pelvic lymphadenectomy or SLN mapping; patients with LSIL on biopsy underwent TCT, HPV, and colposcope 3 months later; if biopsy suggests HSIL and above, perform cone biopsy.
  Interventions: Drug: Camrelizumab; Drug: Cisplatin; Drug: Nab paclitaxel; Procedure: biopsy

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is administered at 200mg, q3w (second and third cycles) before radical surgery
Drug: Cisplatin — 75-80mg/m2, D1-D2，q3w (3 cycles)，intravenous infusion, administered at a rate of 1mg/min.
Drug: Nab paclitaxel — 260 mg/m2，D1，q3w （3 cycles），intravenous infusion, administered over 30min.
Procedure: biopsy — cone biopsy + pelvic lymphadenectomy or Cervical biopsy + pelvic lymphadenectomy

SUMMARY:
This multicenter, prospective clinical trial is designed to enroll PD-L1 expression-positive patients with stage IB1 cervical cancer who desire fertility preservation to undergo neoadjuvant chemotherapy in combination with a PD-1 inhibitor to evaluate the rate of complete pathologic remission, treatment-related adverse events, pregnancy rate, miscarriage rate, preterm birth rate, live birth rate, EFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of stage IB1 cervical cancer after gynecologic examination and MRI evaluation by the investigator (FIGO 2018);
2. Pathologically confirmed diagnosis of cervical squamous cell carcinoma;
3. Transformation zone of TZ1 or TZ2 (IFCPC 2011);
4. Positive PD-L1 expression by preoperative pathology, i.e., Combined Positive Score (CPS) ≥1;
5. Patient age ≥18 years and ≤45 years;
6. ECOG score ≤1;
7. Laboratory tests: white blood cell (WBC) ≥3. 5×109/L, Neutrophil (NEU) ≥1. 5×109/L, platelet (PLT) ≥100×109/L, serum bilirubin ≤1.5 times the upper limit of normal, aminotransferase ≤1.5 times the upper limit of normal, and blood urea nitrogen （BUN) and Cr ≤normal;
8. Have a strong desire to give birth;
9. Willing to sign the informed consent form, including compliance with the requirements and restrictions listed in the informed consent form and program.

Exclusion Criteria:

1. History of infertility, including those with infertility due to tubal or (and) husband;
2. Any active autoimmune disease or history of autoimmune disease requiring systemic treatment, including, but not limited to, autoimmune hepatitis, interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction, asthma requiring bronchodilator intervention;
3. Prior treatment with immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies; known hypersensitivity to any component of the study medication or other monoclonal antibodies;
4. History of human immunodeficiency virus (HIV) infection or known active hepatitis B or C;
5. Use of immunosuppressive drugs or systemic corticosteroid therapy for immunosuppression (>10 mg/day prednisone or equivalent) within 2 weeks prior to study dosing;
6. History of primary malignancy or receipt of chemotherapy or pelvic radiation;
7. Concurrent participation in other clinical trials;
8. Pregnant or breastfeeding female patients; subjects must agree to use effective contraception during study treatment, within 5 months of last use of immune check inhibitors, within 6 months of last use of chemotherapeutic agents, and if there is no confirmation that the lesion has been removed or that the pathology is in remission;
9. Uncontrolled co-morbidities, including but not limited to New York Heart Association (NYHA) class 2 or higher, severe/unstable angina pectoris, myocardial infarction within ≤ 6 months prior to study drug administration, severe arrhythmias requiring medication or intervention; difficult-to-control hypertension; and cerebral vascular accidents or brain disorders within ≤ 6 months prior to study drug administration, or those with adjudicated abnormal behavioral skills; hematologic disorders: coagulation abnormalities (INR > 2. 0, Prothrombin time (PT) > 16s), bleeding tendency, or undergoing thrombolytic or anticoagulant therapy; abnormalities in hepatic or renal development or a history of surgery; and any active infection requiring systemic anti-infective therapy within 14 days prior to the first dose of study drug;
10. Treatment with live or attenuated vaccine within 4 weeks prior to the first dose of study drug; inactivated seasonal influenza virus vaccine is permitted;
11. Patients who have received a previous allogeneic bone marrow or solid organ transplant;
12. Drug and/or alcohol abuse;
13. Patients who, in the opinion of the investigator, are unlikely to comply with the study procedures, restrictions, and requirements may not participate in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | At the end of the patient's treatment, up to 2 years.
  Proportion of patients with no tumor cells on postoperative pathology and negative lymph node metastasis

SECONDARY OUTCOMES:
The negative conversion of HPV | At the end of treatment, up to 2 years.
  Proportion of patients with known HPV infection at screening who are HPV-negative after treatment
Pregnancy rate | Until the end of the 5-year follow-up period, up to 7 years.
  the ratio of the number of women with a successful pregnancy to the total number of women who attempted to become pregnant
Miscarriage rate | Until the end of the 5-year follow-up period, up to 7 years.
  the ratio of miscarriage events that occur during pregnancy in women who are pregnant
Live birth rate | Until the end of the 5-year follow-up period, up to 7 years.
  The live birth rate is the ratio of the number of babies successfully delivered and surviving to the total number of women who attempted pregnancy
Preterm birth rate | Until the end of the 5-year follow-up period, up to 7 years.
  The preterm birth rate is the proportion of babies born at less than 37 weeks of gestation
Adverse Event | during the treatment, up to 5 years.
  Adverse Effects of immunotherapy and chemotherapy
Number of Participants with surgical complications | During and after the surgery, up to 2 years.
  intraoperative bleeding, vascular injuries, bladder injuries, rectal injuries, and ureteral injuries, as defined by the need for suture repair; occlusive nerve injuries, as defined by complete severance; and vascular injuries, as defined by the need to document the site of injury. Postoperative complications included: cervical stenosis, cervical insufficiency, ureteral/bladder/rectal/vaginal fistula, internal hemorrhage, pelvic infection, lymphocyst, lymphatic fistula, lower extremity edema, lower extremity venous thrombosis, urinary retention, nerve injury, and bowel obstruction.
Patient Reported Outcomes (EORTC QLQ-C30) | From enrollment to the end of the 5-year follow-up period. 5 years.
  Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Physical Function Score
Patient Reported Outcomes (EORTC QLQ-CX24) | From enrollment to the end of the 5-year follow-up period. 5 years.
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24) is a questionnaire that rates the symptoms common to women with cervical cancer and evaluates the impact of disease and/or treatments. The 24 items use a 4-point scale (1=not at all to 4=very much) and are classified into 3 multi-item scales, 11 items with symptom experience, 3 items with body image, and 4 items with sexual/ vaginal functioning. The other items of the questionnaire are lymphedema, peripheral neuropathy, menopausal symptom, sexual worry, sexual activity, and sexual enjoyment. The change from baseline in EORTC QLQ-CX24 score will be presented.
Event-free survival (EFS) | Until the end of the 5-year follow-up period, up to 7 years.
  the time between the enrollment and any documented tumor progression, recurrence, or death from any cause; the analysis of EFS includes the results of tumor evaluations during the study treatment and follow-up periods. If a patient had several indicators of progressive disease (PD) or recurrence, the EFS analysis was performed using the indicator that appeared first; PD, recurrence, or death were considered to have reached the study endpoint; patients who were treated with other systemic or antitumor therapies directed at the target lesion of observation were also considered to be in PD; for patients who did not have PD, recurrence, or death at the end of the study, the time when the patient's failure to have a recurrence was last obtained was used as the time to censor the data.
Overall survival (OS) | Until the end of the 5-year follow-up period, up to 7 years.
  the time from the start of enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, Study Chair — Tongji Hospital
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No